CLINICAL TRIAL: NCT06176183
Title: A Comparative Prospective Study of Meniscal Repair Methods in Young Patients With Traumatic Meniscal Tears.
Brief Title: A Comparative Prospective Study of the Arthroscopic Meniscal Repair Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Viktorija Brogaite, Viktorija Brogaite Martinkeniene MD, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/5-1353-825
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Meniscus Tear Caused by a Traumatic Event; Fibrin Clot Augmentation; Meniscal Repair
Keywords: meniscal tear; meniscal repair; fibrin clot; augmentation; arthroscopy; knee; young patients

STUDY DESIGN:
Intervention Model Description: Patients have been randomly assigned into two groups using computerised "randomizer for clinical trial lite". One group of patients has received a standard meniscus suturing technique, whereas another group has experienced the meniscus suturing treatment with an additional fibrin clot approach
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I of patients (Other): Individuals who undergo the conventional arthroscopic meniscus repair procedure
  Interventions: Procedure: Arthroscopic meniscus repair
- Cohort II of patients (Other): Patients who receive the supplementary fibrin clot augmentation during the arthroscopic meniscus repair operation.
  Interventions: Procedure: Arthroscopic meniscus repair

INTERVENTIONS:
Procedure: Arthroscopic meniscus repair — A traditional two-portal arthroscopic approach is utilized. The meniscal edges are examined using a probe, and any meniscal tears that are not stable are evaluated for potential repair. For meniscus repair, sutures have been made using the "all-inside" or "outside-inside" and "inside-outside" techniques.
  If the procedure involving the addition of a fibrin clot is being carried out, a volume of approximately 60 milliliters of blood is taken and thereafter transferred into a basin. An assistant is able to stir the blood using a glass syringe for approximately fifteen minutes to ensure sufficient coagulation surrounding the syringe. After a sufficient clot has developed at the end of the syringe, a grasper is used to insert the clot through the anterolateral arthroscopy portal. The meniscal sutures are intentionally loosened to accommodate the clot in the meniscus, ensuring optimal contact with the lesion. Subsequently, the sutures are fastened and knotted.
  Other Names: Arthroscopic meniscus repair with fibrin clot augmentation

SUMMARY:
Performing arthroscopic meniscus repair following a traumatic meniscus tear as an alternative to a meniscectomy is now an acceptable choice. Preserving meniscus tissues is crucial due to the significant role they play as an essential part of the knee joint. It is essential to comprehend the additional tools that can impact the recovery of the meniscus after suturing. Patients have been randomly assigned into two groups using the computer "www.randomiser.org," and the treatment outcomes were compared after one year. One group of patients has received a standard meniscus suturing technique, whereas another group has experienced the meniscus suturing treatment with an additional fibrin clot approach. Data pertaining to demographics, clinical characteristics, radiological findings, and survey responses have been carefully collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who provide consent to participate in the study, including patients and their care providers. The inclusion criteria for this study are as follows: being under the age of 19, having a traumatic isolated full-thickness meniscal tear longer than 1cm that has been confirmed by both preoperative MRI and arthroscopy, and not having undergone any previous surgery on the affected knee.

Exclusion Criteria:

* This investigation excludes patients with developmental disabilities who are unable to read or interpret in their native language.

Ages: 0 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Pediatric International Documentation Committee Subjective (Pedi-IKDC) Knee Form. | before treatment, after 12 months and 24 months following treatment
  Pedi-IKDC is used to measure knee-related symptoms, function, and sports activity among children. The questionnaire consists of 13 items, each of which is scored using one of three rating systems: a range of 0 to 10 for items 2, 3, 12, and 13, a range of 0 to 4 for items 1, 4, 5, 6, 9, and 10, and a range of 0 to 1 for items 7 and 8. The 11th item consists of nine subquestions, each of which can be scored from 0 to 4. The overall score value is calculated by adding only the responses to 12 items and dividing the total by 92 (the highest number of points attainable). The score runs from 0 (worst case scenario) to 100 (best case scenario). The Pedi-IKDC has been proven to be a valid, trustworthy, and responsive questionnaire in a paediatric population with varied knee disorders, especially ligament and meniscal injuries, joint instability, and other disorders
Lysholm knee scale | before treatment, after 12 months and 24 months following treatment
  Lysholm knee scoring scale has been proven to be suitable for a variety of knee pathologies and also for the adolescent population. The scale comprises eight items. Higher values of the score indicate better functioning of the knee. (range from 0 to 100).
Health-related paediatric quality of life (PedsQL) | before treatment, after 12 months and 24 months following treatment
  PedsQL is a generic score, which estimates the quality of life of paediatric patients. The questionnaire consists of four domains with 23 questions: the general physical functioning, emotional, social, and functioning at school domains

SECONDARY OUTCOMES:
Clinical evaluation at 12 and 24 months postoperatively. The clinical assessment involves evaluating of pain, swelling and estimating and comparing the range of motion of the knee with the contralateral side. | 12 and 24 months postoperatively.
  All patients are evaluated
magnetic resonance imaging (MRI scan) of the knee | before treatment, after 12 months and 24 months following treatment
  1.5T MRI system. Four main diagnostic sequences were analyzed, including sagittal proton density fast spin echo (PD FS-Sag), sagittal T2-weighted fast spin echo (T2W-Sag), coronal proton density fast spin echo with fat saturation (PD FS-Cor), and coronal T2-weighted fast spin echo with fat saturation (T2W-Cor). Signal changes on MRI are graded using Stoller and Crues' 3-stage classification. Grade 0 was defined as a normal meniscus; the meniscus demonstrates low signal intensity in the images. Grade 1 is described as an intrameniscal signal with irregular margins that do not connect or communicate with an articular surface. Grade 2 is defined as a linear signal that does not abut or communicate with an articular surface. A linear or complex signal intensity that abuttes or communicates with an articular surface is classified as Grade 3. In summary, grade 3 is deemed unhealed, grade 2 as partially healed, and grade 1 as fully healed due to MRI assessment.
Revision rates (secondary arthroscopies) | 12 and 24 month following primary surgery
  secondary arthroscopies (revision) at 12 and 24 month following primary surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Lithuania (2):
  - Vilnius University, Medical faculty, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius

IPD SHARING:
Plan to Share IPD: No
As per the study protocol, the IPD has no intention of disclosing the information to third parties or other researchers. In accordance with the data analysis and verification process, the main author of the research could be requested for the provision of anonymized data.